CLINICAL TRIAL: NCT00342693
Title: Thyroid Abnormalities Associated With Protracted Childhood I-131 Exposure From Atmospheric Emissions From the Mayak Nuclear Plant in Russia
Brief Title: Thyroid Abnormalities Associated With Exposure to Atmospheric Emissions of Radioactive Iodine
Status: Terminated | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906103; 06-C-N103
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2013-09-03

CONDITIONS: Thyroid Abnormalities
Keywords: Radiation; Screening; Cancer; Nodules; Nuclear; Thyroid Screening; Thyroid Gland
MeSH Terms: conditions — Thyroid Diseases; Neoplasms

SUMMARY:
Background:

* An inadequate filtering system at the Mayak nuclear weapons production facility in Ozyorsk, Russia, allowed the release of various radioactive materials, particularly I-131 (radioactive iodine) into the city's atmosphere during the 1950s.
* A recent pilot study found a higher prevalence of thyroid nodules in Ozyorsk residents who were exposed to the radiation in childhood during years of heavy atmospheric emissions (1952-1953) than in children exposed in later years (between 1967 and 1991) when there were almost no radioactive releases.
* Understanding the role of I-131 in the development of thyroid disease is important because I-131 is commonly used in medicine (e.g., to treat hyperthyroidism and thyroid cancer and to diagnose thyroid disease), and it is the major source of thyroid gland exposure in fallout from atomic bomb explosions, nuclear power plant accidents, and atmospheric venting from plutonium manufacturing facilities.

Objectives:

-To expand the pilot study to include 350 Ozyorsk residents who were exposed in childhood to moderate levels of radiation in order to evaluate thyroid disease in relation to the dose of I-131 exposure.

Eligibility:

-People who were born and living in Ozyorsk, Russia between 1954 and 1955, the period of mild radioactive releases from the Mayak nuclear weapons plant.

Design:

* Participants' thyroid gland and structure are examined with an ultrasound examination and blood tests.
* Participants with a possible thyroid gland disorder are referred to specialists for additional diagnostic procedures.

DETAILED DESCRIPTION:
We plan to expand a completed pilot study that evaluated the prevalence of thyroid abnormalities in relation to childhood exposure to atmospheric emissions of radioactive iodines from the Mayak Nuclear Weapons Plant in Ozyorsk, Russia. The pilot study population was composed of a defined cohort of approximately 900 Ozyorsk residents who were born between January 1, 1952 and December 31, 1953. The exposed population was comprised of persons who lived in Ozyorsk during the years of heavy atmospheric releases (1952-1953). Members of the nonexposed group moved to Ozyorsk between 1967 and 1991, i.e. when there were almost no radioactive releases. Results from the pilot study suggest an elevated prevalence of thyroid nodules in the exposed population. Given the positive results from the pilot study and the US Department of Energy's (DOE) decision to fund a dose reconstruction project for the Ozyorsk population, we intend to expand the study to include an additional 350 people born and living in Ozyorsk between 1954 and 1955, i.e. exposed to moderate levels of radiation .

Methods similar to those used in the pilot study will be used in the expanded study. Members of the study population will be invited to participate in a special thyroid screening protocol when they come for their annual routine medical examination at the Ozyorsk automated dispensary system (ASDOC). The thyroid gland is clinically examined by two ASDOC physicians specifically trained in thyroid palpation. Thyroid abnormalities will be detected based on physical examinations, assessment of TSH levels, and ultrasound imaging. Biochemical laboratory tests, including Free T(4), and anti-thyroperoxidase antibodies will be assayed as necessary. Patients are sent to a consulting endocrinologist if the palpation, ultrasound or laboratory findings suggest a thyroid disorder. Fine needle aspiration (FNA) biopsy is performed when a tumor is suspected. Although the FNA is not be done as part of the study research, but rather as part of the regular Ozyorsk medical system, the results will be given to the study staff to help make diagnostic decisions. Patients with complicated thyroid disease will be referred to an experienced consulting thyroid specialist. Patients with diagnosed thyroid disease are treated within the regular medical system in Ozyorsk.

ELIGIBILITY:
* Eligibility Criteria:

Currently living and working in Ozyorsk, Russian Federation

Born and living in Ozyorsk between January 1954 and December 1955

Ages: 51 Years to 52 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2006-02-21; Study Completion 2013-09-03

CONTACTS AND LOCATIONS:
Overall Officials: Martha Linet, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Astakhova LN, Anspaugh LR, Beebe GW, Bouville A, Drozdovitch VV, Garber V, Gavrilin YI, Khrouch VT, Kuvshinnikov AV, Kuzmenkov YN, Minenko VP, Moschik KV, Nalivko AS, Robbins J, Shemiakina EV, Shinkarev S, Tochitskaya SI, Waclawiw MA. Chernobyl-related thyroid cancer in children of Belarus: a case-control study. Radiat Res. 1998 Sep;150(3):349-56. PMID 9728663
- [Background] Cardis E, Kesminiene A, Ivanov V, Malakhova I, Shibata Y, Khrouch V, Drozdovitch V, Maceika E, Zvonova I, Vlassov O, Bouville A, Goulko G, Hoshi M, Abrosimov A, Anoshko J, Astakhova L, Chekin S, Demidchik E, Galanti R, Ito M, Korobova E, Lushnikov E, Maksioutov M, Masyakin V, Nerovnia A, Parshin V, Parshkov E, Piliptsevich N, Pinchera A, Polyakov S, Shabeka N, Suonio E, Tenet V, Tsyb A, Yamashita S, Williams D. Risk of thyroid cancer after exposure to 131I in childhood. J Natl Cancer Inst. 2005 May 18;97(10):724-32. doi: 10.1093/jnci/dji129. PMID 15900042
- [Background] Davis S, Stepanenko V, Rivkind N, Kopecky KJ, Voilleque P, Shakhtarin V, Parshkov E, Kulikov S, Lushnikov E, Abrosimov A, Troshin V, Romanova G, Doroschenko V, Proshin A, Tsyb A. Risk of thyroid cancer in the Bryansk Oblast of the Russian Federation after the Chernobyl Power Station accident. Radiat Res. 2004 Sep;162(3):241-8. doi: 10.1667/rr3233. PMID 15332999